CLINICAL TRIAL: NCT06913933
Title: A Two-Arm, Parallel-Group Randomized Controlled Trial Comparing Static Progressive Splinting Versus Dynamic Splinting for Improving Wrist PROM/AROM in Patients With Persistent Post-DRF Stiffness
Brief Title: Static vs. Dynamic Progressive Splinting for Persistent Wrist Stiffness After DRF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al Hayah University In Cairo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPDS2025-03
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Distal Radius Fractures
MeSH Terms: conditions — Wrist Fractures | interventions — Splints

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two parallel arms. One arm will receive a static progressive splint, and the other a dynamic splint, each used in addition to a weekly supervised therapy session. The splints are used to address persistent ROM limitations after conventional therapy has plateaued.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static Progressive Splinting Group (SPSG) (Experimental): Participants in this group receive static progressive splinting using a commercial splint that allows incremental adjustment through a turnbuckle design. This splint is used to gradually increase wrist extension and/or flexion, tailored to the patient's stiffness pattern, alongside a once-weekly supervised therapy session.
  Interventions: Behavioral: Static Progressive Splinting for Persistent Wrist Stiffness
- Dynamic Splinting Group (DSG) (Experimental): Participants in this group receive dynamic splinting using a commercial device equipped with elastic tension (spring-loaded) that provides a constant dynamic stretch to the wrist. This intervention is delivered alongside a weekly supervised therapy session.
  Interventions: Behavioral: Dynamic Splinting for Persistent Wrist Stiffness

INTERVENTIONS:
Behavioral: Static Progressive Splinting for Persistent Wrist Stiffness — A commercially available static progressive splint with a turnbuckle mechanism allowing fine-tuned adjustments in wrist flexion and extension.
  Instructional materials for home use including written guidelines and an adjustment log.
  Arms: Static Progressive Splinting Group (SPSG)
Behavioral: Dynamic Splinting for Persistent Wrist Stiffness — Materials:
  A commercially available dynamic (spring-loaded) splint designed for the wrist. An instructional manual and daily usage log for participants.
  Arms: Dynamic Splinting Group (DSG)

SUMMARY:
This randomized controlled trial will compare the effectiveness of static progressive splinting versus dynamic splinting for treating persistent wrist stiffness in adults ≥18 years old at least 8 weeks post distal radius fracture (DRF) injury. Both splinting modalities are provided as an adjunct to one weekly supervised therapy session over a 6-week period. The primary outcomes are wrist active and passive range of motion (AROM/PROM) measured using goniometry, with secondary outcomes including patient-reported wrist function (PRWE), overall satisfaction, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years or older. At least 8 weeks post distal radius fracture (operative or nonoperative) who have completed standard rehabilitation.

Demonstrated persistent wrist stiffness with ≤50% of contralateral wrist extension or flexion.

Capable of providing written informed consent and complying with study procedures

Exclusion Criteria:

Presence of complex regional pain syndrome (CRPS) or active fracture healing issues.

History of significant wrist pathology unrelated to the DRF. Uncontrolled medical conditions that would interfere with splint application or therapy.

Known skin conditions or allergies that preclude orthosis use. Inability or unwillingness to adhere to the intervention protocol or follow-up schedule.

Pregnant or breastfeeding individuals.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-17 (Estimated); Primary Completion 2026-04-17 (Estimated); Study Completion 2026-04-17 (Estimated)

PRIMARY OUTCOMES:
Wrist Active and Passive Range of Motion (AROM/PROM) | Assessed at baseline, 6 weeks (post-intervention), and 3 months follow-up.
  Measured using a standard goniometer, improvements in wrist flexion and extension (in degrees) are the primary indicators of treatment efficacy.

SECONDARY OUTCOMES:
Patient-Rated Wrist Evaluation (PRWE) | Assessed at baseline and at 6 weeks post-intervention.
  The PRWE questionnaire assesses wrist pain and disability, with lower scores indicating better functional status.
Patient Satisfaction | Collected at 6 weeks and 3 months post-intervention.
  A standardized satisfaction survey measuring patients' perceived improvement and overall satisfaction with the orthotic intervention.
Incidence of Adverse Events | Continuously monitored from baseline to the 3-month follow-up.
  Incidence and severity of adverse events such as skin breakdown, discomfort, or pain (≥4/10) associated with splint usage.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Al Hayah University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No